CLINICAL TRIAL: NCT05802602
Title: Comparison of Porcine Collagen Membrane and Bovine Collagen Wound Dressing in Human Extraction Sites With DFDBA Graft: A Randomized Controlled Trial
Brief Title: Porcine Membrane vs Bovine Wound Dressing in Human Tooth Extraction Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0145-23-FB
Record Dates: First submitted 2023-03-02; First posted 2023-04-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-05

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Porcine Collagen Membrane (Experimental): Atraumatic tooth extraction with porcine collagen membrane placement
  Interventions: Device: Porcine Collagen Membrane
- Bovine Collagen Dressing (Active Comparator): Atraumatic tooth extraction with bovine collagen dressing placement
  Interventions: Device: Bovine Collagen Dressing

INTERVENTIONS:
Device: Porcine Collagen Membrane — Atraumatic tooth extraction with porcine collagen membrane placement
  Other Names: Mucograft
  Arms: Porcine Collagen Membrane
Device: Bovine Collagen Dressing — Atraumatic tooth extraction with bovine collagen dressing placement
  Other Names: Heliplug
  Arms: Bovine Collagen Dressing

SUMMARY:
The purpose of this study is to compare porcine collagen membrane and bovine collagen wound dressing in human tooth extraction sites. The outcomes measured will be soft tissue thickness changes as well as bone density changes.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of a porcine collagen membrane to a bovine collagen wound dressing for atraumatic extractions. These are both commonly used as a barrier and containment material over atraumatic extraction sites that are grafted for future implant placement. The study will include nonsmoking adults aged 18-65 requiring premolar or anterior tooth extraction and graft procedures, who are in good general health and willing to provide informed consent. Exclusion criteria include a history of radiation therapy or bisphosphonate use, pregnancy or breastfeeding, systemic conditions that affect bone healing, contraindications to dental implants, and inability to attend follow-up visits. The study will be a double-blind randomized controlled trial involving 24 patients who will be assigned to two groups. Prior to tooth extraction, baseline data will be collected; including gingival crevicular fluid (GCF) sampling, and a limited field Cone Beam Computed Tomography (CBCT) radiograph. A reference digital scan will be taken to measure volumetric changes in soft tissue. Routine, atraumatic extraction of the tooth under local anesthetic will be performed. Following extraction, hydrated AllOss 50/50 DFDBA:FDBA (demineralized freeze-dried bone allograft:freeze-dried bone allograft) bone particulate will be condensed following a routine protocol. One group will receive Mucograft Seal over the graft, and the other group will receive Integra HeliPlug. Patients will be seen at a standard 2-week follow up to remove sutures, have a GCF sampling at the adjacent teeth and take another digital scan. Patients will be seen for an additional 6-week follow up to take a small (2mm) incisional biopsy for histological analysis. Another digital scan and GCF sampling will be taken. Final evaluation will be 3 months post-extraction and will include a localized CBCT evaluation for implant planning and another measure of soft tissue changes with a digital scan. At the time of implant surgery, the core of bone removed during osteotomy will be histologically analyzed for percentage of vital bone. Adverse events will also be recorded at each visit. The primary outcome measure will be the histological composition of tissue at 6 weeks and volumetric tissue changes. The secondary outcome measures will be bone density changes on the post-operative CBCT and inflammatory bio-markers present at baseline, 2-weeks via GCF sampling.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Aged 19-65
* Requiring premolar or anterior tooth extraction and graft procedures
* Good general health
* Willing to provide informed consent.

Exclusion Criteria:

* History of radiation therapy or bisphosphonate use
* Pregnancy or breastfeeding
* Systemic conditions that affect bone healing
* Contraindications to dental implants
* Inability to attend follow-up visits.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-04-16 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Soft Tissue Thickness in mm | 6 weeks
  Soft tissue biopsy to determine tissue thickness, measured in mm

SECONDARY OUTCOMES:
Bone Density Measurements | Baseline, 3 Months
  Bone density measurements to assess vital bone, bone tissue that retains living cells and a blood supply, at the extraction site CBCT measurement of bone density at baseline and three months, measured in Hounsfield units
Interleukin-1beta | Baseline, 2 Weeks & 6 Weeks
  Interleukin-1beta (IL-1β), a pro-inflammatory cytokine primarily produced by immune cells and measured in pg/mL, will be assessed from gingival crevicular fluid (GCF) samples around the extraction site taken at baseline, 2 weeks and 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, MS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT05802602/Prot_000.pdf
  • Informed Consent Form (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT05802602/ICF_001.pdf